CLINICAL TRIAL: NCT01238887
Title: Investigations of Botanicals on Food Intake, Satiety, Weight Loss, and Oxidative Stress
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Some capsules used in this study were been found to be cracked and leaking.
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 001; K23AT004251 (NIH)
Record Dates: First submitted 2010-08-06; First posted 2010-11-11 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Oxidative Stress
Keywords: Satiety; Food Intake; Weight Loss; Oxidative Stress; botanicals; Garcinia Cambogia-derived hydroxycitric acid
MeSH Terms: conditions — Obesity; Weight Loss | interventions — hydroxycitric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- microcrystalline cellulose (Placebo Comparator)
  Interventions: Dietary Supplement: Microcrystalline Cellulose placebo pill
- Hydroxycitric acid (Active Comparator): 2800 mg divided in three doses per day
  Interventions: Dietary Supplement: Garcinia cambogia-derived hydroxycitric acid (2800 mg/day); Dietary Supplement: Garcinia Cambogia derived Hydroxycitric Acid
- Hydroxycitric Acid (Active Comparator): 5400 mg divided into three doses per day
  Interventions: Dietary Supplement: Garcinia cambogia-derived hydroxycitric acid (2800 mg/day); Dietary Supplement: Garcinia Cambogia derived Hydroxycitric Acid

INTERVENTIONS:
Dietary Supplement: Microcrystalline Cellulose placebo pill — Participants will be given gelatin capsules containing the placebo (microcrystaline cellulose) and will be instructed to consume four capsules three times daily (30 minutes before breakfast, lunch, and dinner) with a glass of water. This will equal 3000 mg/day of the placebo contents. Participants will be instructed to follow this dosing regimen throughout the six week treatment period.
  Arms: microcrystalline cellulose
Dietary Supplement: Garcinia cambogia-derived hydroxycitric acid (2800 mg/day) — The hydroxycitric acid treatment is derived from garcinia cambogia and is provided by the company, Glykon Technologies. In this condition, participants will receive HCA at a dosage of 2,800 mg/day in the form of gelatin capsules. Participants will be instructed to consume four capsules three times daily (30 minutes before breakfast, lunch, and dinner) with a glass of water. Participants will be instructed to follow this dosing regimen throughout the six week treatment period.
  Other Names: Hydroxycitric Acid (HCA)
  Arms: Hydroxycitric Acid; Hydroxycitric acid
Dietary Supplement: Garcinia Cambogia derived Hydroxycitric Acid — The hydroxycitric acid treatment is derived from garcinia cambogia and is provided by the company, Glykon Technologies. In this condition, participants will receive HCA at a dosage of 5,400 mg/day in the form of gelatin capsules. Participants will be instructed to consume four capsules three times daily (30 minutes before breakfast, lunch, and dinner) with a glass of water. Participants will be instructed to follow this dosing regimen throughout the six week treatment period.
  Other Names: Hydroxycitric Acid (HCA)
  Arms: Hydroxycitric Acid; Hydroxycitric acid

SUMMARY:
Despite widespread efforts to improve the treatment of obesity, only limited progress has been made. Calorie restriction (CR) has consistently been shown to produce weight loss, as well as delay the onset of age-related diseases, in numerous species. Most overweight individuals, however, are unable to sustain CR induced weight losses, possibly due to internal feedback systems that signal the body to increase food intake or decrease energy expenditure in response to weight loss. Novel treatment approaches are thus urgently needed that can assist overweight individuals in adhering to a CR regimen over the long-term.

Botanicals represent an important and underexplored source of potential new therapies that may facilitate CR. In particular, one promising botanical that may reduce food intake and body weight by affecting neuroendocrine pathways related to satiety is Garcinia Cambogia (Garcinia Cambogia Desr.)-derived (-)-hydroxycitric acid. This compound has been found to facilitate weight loss in a number of studies. To date, few studies have directly tested the effect that this botanical on food intake in humans, its mechanism of action, or its effect on oxidative stress levels; thus rigorous scientific studies on this compounds need to be conducted. A double-blind, placebo-controlled crossover study will be conducted to explore the role that two different doses of this botanical compound have on food intake, satiety, weight loss, and oxidative stress levels. It is hypothesized that compared to placebo, both doses of Garcinia Cambogia (hydroxycitric acid) will reduce food intake, increase satiety, decrease weight, and reduce oxidative stress levels.

ELIGIBILITY:
Inclusion Criteria:

1. healthy individual with normal blood chemistries and platelet counts who has not been diagnosed with diabetes, cardiovascular illness, or other chronic diseases
2. 50 to 70 years of age
3. body mass index between 25 and 39.9 kg/m2
4. for females, post-menopausal (i.e., no menstrual cycle for > one year).

Exclusion Criteria:

1. Potential participants will be excluded if their scores on the dietary restraint, disinhibition, and perceived hunger scales of the Eating Inventory are high (>14)
2. Participants who report smoking cigarettes will be excluded because of the effects of nicotine upon taste and appetite
3. Participants who have a diagnosable eating disorder will also be excluded since intentional restriction of eating and binge eating/overeating could increase the variability of the data
4. Participants will be excluded if they are taking anti-depressant medications, anti-psychotic medications, or any medications, botanicals, or other products that may potentially influence appetite, hunger, and/or satiety
5. Participants will be excluded if they report alcohol or substance abuse within 6 months or consumption of >14 alcohol drinks/week
6. Participants will also be excluded if they report any allergies to the foods used in the study
7. Volunteers will also be ineligible if they have significant medical conditions (e.g., history or clinical manifestation of cardiovascular disease, diabetes, cholelithiasis, liver or renal disease, or cancer)

   * abnormal laboratory markers (e.g., renal or liver abnormalities, elevated potassium levels or hemoglobin and hematocrit below the lower limit of normal)
   * psychiatric or behavioral problems (e.g., eating disorders or a history of drug and alcohol abuse)
   * concomitant medications (e.g., steroids)
8. Volunteers will be screened out if they are unwilling or unable to adhere to different supplement regimens over an eight month period.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Food Intake (kcal/day) | Measured every six weeks over a 30 week period
  Participant food intake will be measured at each meal of every test meal day, once at breakfast, lunch, and dinner. Test meal days occur at the baseline visit, after six weeks of the the first condition (week 6), after the following six week wash out period (week 12), after the following six weeks of the second condition (week 18), after the following six week wash out period (week 24), and after the six weeks of the third and final condition (week 30). Conditions include both the doses of the treatment and the placebo dose as well.

SECONDARY OUTCOMES:
Satiety | Measured every six weeks over a 30 week period
  Participants will provide satiety ratings throughout the test meal day. Test meal days occur at the baseline visit, after six weeks of the the first condition (week 6), after the following six week wash out period (week 12), after the following six weeks of the second condition (week 18), after the following six week wash out period (week 24), and after the six weeks of the third and final condition (week 30).
Body Weight | Every six weeks over a 30 week period
  Fasting body weights will be taken at each of the test meal visits. Test meal days occur at the baseline visit, after six weeks of the the first condition (week 6), after the following six week wash out period (week 12), after the following six weeks of the second condition (week 18), after the following six week wash out period (week 24), and after the six weeks of the third and final condition (week 30).
Oxidative Stress | Every Six weeks for 30 weeks
  Fasting blood draws will be taken at each of the test meal visits. Test meal days occur at the baseline visit, after six weeks of the the first condition (week 6), after the following six week wash out period (week 12), after the following six weeks of the second condition (week 18), after the following six week wash out period (week 24), and after the six weeks of the third and final condition (week 30).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anton, Ph.D., Principal Investigator — University of Florida, Department of Aging and Geriatric Research
Locations (1):
- University of Florida General Clinical Research Center (GCRC), Gainesville, Florida, United States

REFERENCES:
- [Background] Kenchaiah S, Evans JC, Levy D, Wilson PW, Benjamin EJ, Larson MG, Kannel WB, Vasan RS. Obesity and the risk of heart failure. N Engl J Med. 2002 Aug 1;347(5):305-13. doi: 10.1056/NEJMoa020245. PMID 12151467
- [Derived] Anton SD, Shuster J, Leeuwenburgh C. Investigations of botanicals on food intake, satiety, weight loss and oxidative stress: study protocol of a double-blind, placebo-controlled, crossover study. Zhong Xi Yi Jie He Xue Bao. 2011 Nov;9(11):1190-8. doi: 10.3736/jcim20111106. PMID 22088584